CLINICAL TRIAL: NCT06471374
Title: Pathophysiology of Circadian Rhythm Delayed Sleep Wake Phase Disorder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Boulder (Other)
Collaborators: Northwestern University (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Kenneth Wright, Professor, University of Colorado, Boulder
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 23-0285; 1R01HL159647-01 (NIH)
Record Dates: First submitted 2024-06-18; First posted 2024-06-24 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2024-06

CONDITIONS: Delayed Sleep Phase Syndrome; Delayed Sleep Phase
MeSH Terms: conditions — Sleep Disorders, Circadian Rhythm

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Assessment (Experimental): Circadian rhythms and light sensitivity
  Interventions: Behavioral: Circadian rhythm assessment; Behavioral: Light sensitivity assessment

INTERVENTIONS:
Behavioral: Circadian rhythm assessment — Participants will arrive approximately 8 hours before participant's scheduled bedtime to practice ability to think testing and a 9-hour sleep study. Participants will live in the laboratory for approximately 66 hours (2.75 days). Upon awakening in the morning, participants will start a routine of up to 39 hours of wakefulness, under bedrest conditions. Saliva will be sampled frequently and blood will be drawn 3 times. Reaction time, ability to think, and subjective rating tests will be performed frequently. Participants will be provided scheduled bathroom breaks when participants will use a commode next to the bed. Outside these scheduled bathroom breaks, participants will be provided a bedpan to use to go to the bathroom. At the end of the research procedures for Visit 4 participants will be given a recovery sleep opportunity and be discharged from the lab in the morning near participant's typical waketime.
Behavioral: Light sensitivity assessment — Participants will arrive in the afternoon to practice ability to think testing and a 9-hour sleep study. Participants will live in the laboratory for approximately 48 hours (2 days). Upon awakening in the morning, participants will be exposed to dim candlelight and then later in the day alternating intensities of dim and room light when we keep participants awake for up to 23 hours (We will ask participants to remain in bed seated for ~12.5 hours). Saliva will be sampled frequently. Reaction time, ability to think, and subjective rating tests will be performed frequently. Participants will then have a second 9-hour sleep opportunity.

SUMMARY:
The goal of this study is to understand factors that contribute to delayed sleep wake phase disorder (DSWPD). The investigators will examine whether patients with DSWPD exhibit alterations in circadian rhythms and sensitivity to light compared to healthy controls. The investigators will also test a new method of predicting circadian rhythms form a blood sample.

DETAILED DESCRIPTION:
* The research parts of the study are 6.5 weeks long and the study, including screening visits, involves 6 in-person visits to the Boulder campus.
* If participants qualify for the study and choose to participate, there will be two visits where participants will pick up research equipment to wear at home for 1-2 weeks of ambulatory monitoring before being studied in the laboratory. The first ambulatory monitoring session is for 2 weeks and the second is one week.

  * On the first ambulatory monitoring session the investigators will have participants answer questions about participant's mood and cognition.
  * On both ambulatory monitoring sessions, the investigators will also ask participants to wear a blood sugar monitor and track the timing of when participants eat using a phone app. The investigators will also have participants wear a wrist worn sleep and light monitor plus a daily sleep log and Google form of when participants go to bed and wake up.
* Next will be a visit where participants will spend 66 hours (2.75 days) in the laboratory.

  * While living in the lab, participants will not be aware of the time of day (e.g., no clocks, internet, cell phones), and the investigators will schedule participant's activities.
  * The investigators will ask participants to remain seated in bed and awake for up to ~39 hours, with the head of the bed raised. Participants will be studied under dim light similar to candlelight.
  * The investigators will frequently take saliva samples for more than 24 hours when the investigators will ask participants to stay awake. The investigators will also take four blood samples.
  * The investigators will also ask participants to perform reaction time tests, tests of participant's ability to think, and to complete ratings of how participants feel multiple times each day that participants are in the lab.
  * The investigators will also record participant's brain wave activity, muscle activity, eye movements, and heart rate when participants stay awake and during ~9h sleep opportunities.
* The investigators will then ask participants to sleep normally at home for ~2 weeks, followed by 1 week of ambulatory monitoring.
* Finally, there will be a visit where participants will spend 48 hours (2 days) in the laboratory.

  * While living in the lab, participants will not be aware of the time of day (e.g., no clocks, internet, cell phones) and the investigators will schedule participant's activities.
  * The investigators will expose participants to different light levels (dim light similar to candlelight and typical room light).
  * The investigators will frequently take saliva samples.
  * The investigators will also ask participants to perform reaction time tests, tests of participant's ability to think, and to complete ratings of how participants feel multiple times each day that participants are in the lab.
  * The investigators will also record participant's brain wave activity, muscle activity, eye movements, and heart rate when participants are awake and while participants sleep.

ELIGIBILITY:
Inclusion Criteria:

* Delayed sleep wake phase disorder diagnosis
* Altitude history: currently residing at Denver altitude or higher
* BMI normal to moderately overweight

Exclusion Criteria:

* Recent medical condition
* Psychiatric disorder
* Sleep disorder
* Medication use

Ages: 16 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 66 (Estimated)
Dates: Start 2024-04-02 (Actual); Primary Completion 2028-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Core body temperature | Continuously for 1. up to 39 and 2. 23 hours
  Body temperature measured with a pill
Glucose | Continuously for 1. up to 39 and 2. 23 hours
  Blood sugar levels
Subjective sleepiness | Every 2 hours
  Self reported sleepiness
Psychomotor vigilance | Every 2 hours
  Attention/Vigilance performance

SECONDARY OUTCOMES:
Skin temperature | Continuously for 1. up to 39 and 2. 23 hours
  skin body temperature
Melatonin | Hourly for 1. up to 39 hours and 2. every 20 minutes
  Melatonin levels in saliva

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Wright, PhD, Principal Investigator — University of Colorado, Boulder
Locations (2):
- United States (2):
  - University of Colorado, Boulder, Colorado
  - Northwestern University, Chicago, Illinois